CLINICAL TRIAL: NCT02414217
Title: Intervention to Enhance Numeracy in Diabetes
Brief Title: Intervention to Enhance Numeracy in Diabetes (IntEND)
Acronym: IntEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0229
Record Dates: First submitted 2015-04-02; First posted 2015-04-10 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Diabetes
Keywords: numeracy; health literacy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Diabetes Numeracy Education (Experimental): Participants randomized to the in-person education group attended four group classes, each addressing a specific set of diabetes self-care skills (i.e., understanding and using blood glucose numbers, counting carbohydrates, taking medications at the right dose and time). So that each class included a stable group of 8 and 16 participants, we ran classes in "cohorts" of 8-16 people. A participant always attended classes with his/her cohort.
  Interventions: Behavioral: In-Person Diabetes Numeracy Education
- Online Diabetes Numeracy Education (Experimental): Participants randomized to the online education group attended a single session, at which he/she completed a computerized education module that addressed understanding blood sugar values and using them to examine the impact of food, exercise, and medicines on blood sugar.
  Interventions: Behavioral: Online Diabetes Numeracy Education
- Control (No Intervention): Participants were given written educational materials about diabetes.

INTERVENTIONS:
Behavioral: In-Person Diabetes Numeracy Education — Participants randomized to the in-person education group attended four group classes, each addressing a specific set of diabetes self-care skills (i.e., understanding and using blood glucose numbers, counting carbohydrates, taking medications at the right dose and time). So that each class included a stable group of 8 and 16 participants, we ran classes in "cohorts" of 8-16 people. A participant always attended classes with his/her cohort.
  Other Names: Intervention to Enhance Numeracy in Diabetes (IntEND)
  Arms: In-Person Diabetes Numeracy Education
Behavioral: Online Diabetes Numeracy Education — Participants randomized to the online education group attended a single session, at which he/she completed a computerized education module that addressed understanding blood sugar values and using them to examine the impact of food, exercise, and medicines on blood sugar.
  Other Names: Electronic Diabetes Numeracy Intervention (e-DNI)
  Arms: Online Diabetes Numeracy Education

SUMMARY:
The objective of this project is to test two interventions designed to improve diabetes-related numeracy. Numeracy is the ability to understand and use numbers. People with diabetes use numbers in a variety of ways in managing their condition (e.g., understanding blood sugar values, counting carbohydrates, taking medications at the right dose and time). As part of this project, the investigators developed and pilot tested two interventions to improve diabetes-related numeracy: (1) a series of in-person education classes and (2) a one-time, online diabetes education class. The investigators will look to see whether participants in the education classes show improvements in their diabetes-related numeracy skills, self-care behavior and attitudes, and clinical outcomes (i.e., body mass index, blood pressure, blood sugar [A1c]).

DETAILED DESCRIPTION:
Sixty-five American Indians with diabetes were enrolled. Each participant was randomly assigned to 1 of 3 study arms: (1) the in-person education group, (2) the online education group, and (3) a control group. The in-person intervention group attended four class sessions addressing numeracy skills used in the management of diabetes (e.g., counting carbohydrates). The online education group completed a single online module providing training on diabetes-related numeracy skills. The control group received written diabetes educational materials. The investigators collected data at baseline, then again immediately after intervention participation (in-person or online classes), and one final time about three months after the conclusion of the intervention. The investigators will conduct analyses to determine if intervention participants experienced positive changes in diabetes numeracy (the primary outcome) as well as several secondary outcome measures following intervention. Secondary outcomes include: diabetes knowledge, self-efficacy, outcome expectancies, readiness to change, self-care behavior, and clinical outcomes (i.e., body mass index, blood pressure, blood sugar [A1c]) . The investigators also will assess whether change in numeracy predicts change in these secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Indian/Alaska Native;
* 18 to 89 years old;
* diabetes diagnosis documented in medical records;
* active patient of the Yakama Indian Health Service.

Exclusion Criteria:

* Does not speak English;
* pregnancy;
* dialysis;
* current cancer treatment;
* blindness;
* active alcohol/substance abuse;
* planning to move out of the area in the next six months.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Objective Diabetes Numeracy from Baseline to ≈6 weeks | ≈6 weeks
  Adapted version of the Diabetes Numeracy Test

SECONDARY OUTCOMES:
Change in Objective Diabetes Numeracy from Baseline to ≈3 months | ≈3 months
  Adapted version of the Diabetes Numeracy Test
Change in Subjective Numeracy from Baseline to ≈6 weeks | ≈6 weeks
  Subjective Numeracy Scale
Change in Subjective Numeracy from Baseline to ≈3 months | ≈3 months
  Subjective Numeracy Scale
Change in Diabetes Knowledge from Baseline to ≈6 weeks | ≈6 weeks
  Adapted version of the Diabetes Knowledge Test
Change in Diabetes Knowledge from Baseline to ≈3 months | ≈3 months
  Adapted version of the Diabetes Knowledge Test
Change in Diabetes Self-Efficacy from Baseline to ≈6 weeks | ≈6 weeks
  Adapted items from existing instruments
Change in Diabetes Self-Efficacy from Baseline to ≈3 months | ≈3 months
  Adapted items from existing instruments
Change in Outcome Expectancies from Baseline to ≈6 weeks | ≈6 weeks
  Adapted items from existing instruments
Change in Outcome Expectancies from Baseline to ≈3 months | ≈3 months
  Adapted items from existing instruments
Change in Readiness to Change from Baseline to ≈6 weeks | ≈6 weeks
  Newly developed items
Change in Readiness to Change from Baseline to ≈3 months | ≈3 months
  Newly developed items
Change in Diabetes Self-Care Behavior from Baseline to ≈6 weeks | ≈6 weeks
  Summary of Diabetes Self-Care Activities Scale plus additional relevant items
Change in Diabetes Self-Care Behavior from Baseline to ≈3 months | ≈3 months
  Summary of Diabetes Self-Care Activities Scale plus additional relevant items
Change in Body Mass Index from Baseline to ≈6 weeks | ≈6 weeks
  Body Mass Index
Change in Body Mass Index from Baseline to ≈3 months | ≈3 months
  Body Mass Index
Change in Blood Pressure from Baseline to ≈6 weeks | ≈6 weeks
  Systolic and Diastolic Blood Pressure
Change in Blood Pressure from Baseline to ≈3 months | ≈3 months
  Systolic and Diastolic Blood Pressure
Change in Glycemic Control from Baseline to ≈3 months | ≈3 months
  Hemoglobin A1c

CONTACTS AND LOCATIONS:
Overall Officials: Angela G. Brega, PhD, Principal Investigator — University of Colorado, Denver